CLINICAL TRIAL: NCT06258447
Title: Randomized Controlled Pivotal Trial of Autologous Bone Marrow Mononuclear Cells Using the CardiAMP Cell Therapy System in Patients With Ischemic Heart Failure II Trial
Brief Title: CardiAMP Heart Failure II Trial for Patients With Ischemic Heart Failure With Reduced Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioCardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05804 (CLIN)
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Intervention Model Description: Controlled study of study treatment consisting of intramyocardial autologous cell injections compared to sham control, both performed in cardiac catheterization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind including study participants and care provider (investigator) conducting outcomes assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study (ABM MNC) Treatment (Experimental): Left ventricular catheterization with treatment consisting of autologous bone marrow mononuclear cells (ABM MNC) processed and delivered using the CardiAMP cell therapy system
  Interventions: Device: Autologous bone marrow mononuclear cells processed / delivered using the CardiAMP cell therapy system
- Control Treatment (Sham Comparator): Left ventricular (diagnostic) catheterization but no administration of ABM MNC
  Interventions: Device: Autologous bone marrow mononuclear cells processed / delivered using the CardiAMP cell therapy system

INTERVENTIONS:
Device: Autologous bone marrow mononuclear cells processed / delivered using the CardiAMP cell therapy system — the ABM MNC is obtained from the study patient via bone marrow aspiration in the hip and processed and delivered using the CardiAMP cell therapy system during the cardiac catheterization.

SUMMARY:
Concentrated autologous bone marrow mononuclear cells (ABM MNC) contain potentially therapeutic cell factors and past studies support therapeutic benefit to patients with cardiac diseases of acute myocardial infarction, ischemia, and heart failure when utilized as this study is designed. The purpose of the study is to determine the safety and efficacy of CardiAMP cell therapy system in patients with ischemic heart failure. It is a prospective, multi-center, randomized, controlled, patient and evaluator-blinded study comparing treatment with the CardiAMP cell therapy system to a control procedure with diagnostic catheterization.

DETAILED DESCRIPTION:
Chronic heart failure is in need of new therapies. Over the past few years, cardiovascular regenerative medicine using bone marrow derived cells has emerged as a new treatment strategy that could have tremendous benefit in treating heart failure and are well supported by recent meta analyses of early clinical data sets. Concentrated autologous bone marrow mononuclear cells (ABM MNC) are the subject of the current study as they are supported by more clinical data than any other cell type described, and contain all of the potentially therapeutic cell factors from studies of selected cells. Study results demonstrate ABM MNC to be safe, and, when delivered intramyocardially as intended in the current study, results consistently support therapeutic benefit to patients with cardiac diseases of acute myocardial infarction, ischemia, and heart failure. The purpose of the study is to determine the safety and efficacy of CardiAMP cell therapy system in patients with ischemic heart failure. It is a prospective, multi-center, randomized, controlled, patient and evaluator-blinded study comparing treatment with the CardiAMP cell therapy system to a control procedure with diagnostic catheterization. The Treatment Group undergoes left ventricular catheterization and is treated with ABM MNC using the CardiAMP cell therapy system. The Control Group has a Control procedure consisting of left ventricular diagnostic catheterization but no introduction of the Helix transendocardial delivery catheter and no administration of ABM MNC.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) Class II or III
* Diagnosis of chronic ischemic left ventricular dysfunction secondary to myocardial infarction (MI) as described in the study protocol.
* Left ventricular ejection fraction >20% and <40%
* On stable evidence-based medical and device therapy for ischemic etiology heart failure per the ACC/AHA Heart Failure guidelines, for at least three (3) months prior to randomization.
* NTproBNP level of >500 pg/ml
* Autologous cell analysis score consistent with study selection assessment

Exclusion Criteria:

* Selected study criteria as defined in the study protocol indicating that patient is not an optimal candidate for cardiac catheterization or intramyocardial delivery of autologous bone marrow mononuclear cells.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | Follow-up duration at endpoint analysis ranges from a minimum of 12 to a maximum of 24 months
  The primary efficacy endpoint is the comparison of a composite score based on a 3-tiered Finkelstein-Schoenfeld (FS) hierarchical analysis. The tiers, starting with the most serious events, would be (1) all cause death, including cardiac death equivalents such as heart transplant or left ventricular assist device placement, ordered by time to event; (2) non-fatal MACCE events (heart failure hospitalization or a worsening heart failure, stroke or MI) ordered by time to event, excluding those deemed procedure related occurring within the first 7 days, and (3) change for quality of life as measured using the Minnesota Living with Heart Failure Questionnaire (MLwHFQ)

SECONDARY OUTCOMES:
First Secondary Endpoint | Baseline through study completion, maximum of two years
  Time to all-cause death, LVAD/heart transplant, or heart failure hospitalization
Second Secondary Endpoint | Baseline through study completion, maximum of two years
  Cumulative heart failure hospitalizations
Third Secondary Endpoint | Baseline through study completion, maximum of two years
  Time to first heart failure hospitalization
Fourth Secondary Endpoint | Baseline to 12 months, 24 months
  Change in quality of life as measured using the MLwHF questionnaire based on a scale of 0-105, with 0 being best.
Fifth Secondary Endpoint | Baseline to 12 months, 24 months
  Change in quality of life as measured using the Kansas City Cardiomyopathy questionnaire (KCCQ), based on a scale of 0-100, with 100 being best
Sixth Secondary Endpoint | Baseline to 12 months, 24 months
  Change in functional capacity as measured using the 6-minute walk test (6MWT)
Seventh Secondary Endpoint | Baseline through study completion, maximum of two years
  Modified Primary Efficacy Endpoint consisting of all-cause death, LVAD/heart transplant, heart failure hospitalizations and worsening heart failure events treated as an outpatient but without a quality-of-life measure

CONTACTS AND LOCATIONS:
Overall Officials: Amish Raval, MD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - Morton Plant Hospital - BayCare, Clearwater, Florida
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Wisconsin-Division of Cardiovascular Medicine, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No plan at this time to make IPD available to other researchers.